CLINICAL TRIAL: NCT04854447
Title: Part-time Versus Full-time Spectacles for Myopia Control (ParMA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: State Scholarships Foundation (Unknown)
Responsible Party: Principal Investigator, Asimina Mataftsi, Associate Professor in Ophthalmology, Paediatric Ophthalmology and Strabismus, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.68/27-02-2019
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Myopia
Keywords: Myopia; Spectacles; Full-time correction; Part-time correction; Childhood
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Part-time myopia correction with single-vision spectacles
  Interventions: Device: Single-Vision Spectacles
- Control Group (Active Comparator): Full-time myopia correction with single-vision spectacles
  Interventions: Device: Single-Vision Spectacles

INTERVENTIONS:
Device: Single-Vision Spectacles — Spectacle correction for myopia treatment

SUMMARY:
The purpose is to assess the effect of part-time compared to full-time spectacle use in juvenile myopia control.

DETAILED DESCRIPTION:
A prospective, randomized, controlled clinical trial was designed for assessing the effect of single-vision spectacles on myopic progression. 30 myopic subjects, aged 6-16 years old, with a spherical equivalent refraction between -0.50D and -6.00D, were recruited. A random number table was used to allocate participants into either a) part-time use of single-vision spectacles, or b) full-time use of single-vision spectacles. Part-time use was for 4-6 hours a day, 7 days a week for a year. Clinical assessment included follow-up at 6 months and at 12 months upon allocation. The primary outcomes were a) change in spherical equivalent refraction (SER) measured by cycloplegic autorefraction, and b) change in axial eye length (AL). The secondary outcomes were a) change in choroidal thickness (ChT), and b) assessment of the subjective tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 16 years old at the time of enrollment.
* Best-corrected visual acuity (BCVA) LogMAR 0.1 or better, in each eye.
* Cycloplegic Autorefraction: Myopia, SER between -0.50D and -6.00D, in each eye. Astigmatism less than or equal to 1.50D, in each eye. Anisometropia less than or equal to 1.50D between the two eyes.
* Absence of any ocular or systemic condition that could influence refractive development, other than myopia.
* Eagerness to participate in this study and receive myopia treatment in a randomized fashion. Availability for at least 1-year follow-up. Subject parent's or guardian's understanding of the protocol and acceptance to participate, providing a signed consent on behalf of the subject.

Exclusion Criteria:

* Presence of strabismus.
* Presence of amblyopia.
* Prematurity (gestational age less than 37 weeks).
* Presence of an ocular condition affecting refraction (ie. cataract, dislocated lens).
* Presence of a systemic condition affecting refraction (ie. Down syndrome, Marfan syndrome).
* Allergy to cyclopentolate. Severe ocular or systemic allergies.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Change in spherical equivalent refractive error (SER), measured using cycloplegic autorefraction. | Baseline to 6-months, and baseline to 12-months.
Change in axial length (AL). | Baseline to 6-months, and baseline to 12-months.

SECONDARY OUTCOMES:
Change in choroidal thickness (ChT). | Baseline to 6-months, and baseline to 12-months.
Subjective tolerance, as assessed using a standardized questionnaire created for the purpose of this study. | Baseline to 12-months.
  This questionnaire is formed by the researchers participating in this study and is aimed at providing a qualitative assessment of the subjective tolerance of included children wearing spectacles. It incorporates 6 questions and is not based on a scale.

CONTACTS AND LOCATIONS:
Locations (1):
- "Papageorgiou" General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasudevan B, Esposito C, Peterson C, Coronado C, Ciuffreda KJ. Under-correction of human myopia--is it myopigenic?: a retrospective analysis of clinical refraction data. J Optom. 2014 Jul-Sep;7(3):147-52. doi: 10.1016/j.optom.2013.12.007. Epub 2014 May 10. PMID 25000870
- [Background] Sun YY, Li SM, Li SY, Kang MT, Liu LR, Meng B, Zhang FJ, Millodot M, Wang N. Effect of uncorrection versus full correction on myopia progression in 12-year-old children. Graefes Arch Clin Exp Ophthalmol. 2017 Jan;255(1):189-195. doi: 10.1007/s00417-016-3529-1. Epub 2016 Oct 29. PMID 27796670
- [Background] Logan NS, Wolffsohn JS. Role of un-correction, under-correction and over-correction of myopia as a strategy for slowing myopic progression. Clin Exp Optom. 2020 Mar;103(2):133-137. doi: 10.1111/cxo.12978. Epub 2019 Dec 18. PMID 31854025